CLINICAL TRIAL: NCT00449852
Title: An Interactive, Voice Response-Mediated, Follow-up and Triage System for Smoking Cessation in Smokers With Coronary Heart Disease
Brief Title: Interactive Voice Response Telephone Technology for the Treatment of Smoking in Patients With Heart Disease
Acronym: IVR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other)
Responsible Party: Robert Reid PhD MBA, University of Ottawa Heart Institute
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: NA 5845
Record Dates: First submitted 2007-03-19; First posted 2007-03-21 (Estimated); Last update posted 2011-04-29 (Estimated); Status verified 2011-04

CONDITIONS: Coronary Artery Disease
Keywords: Randomized Control Trial; Smoking Cessation; Secondary Prevention; Rehabilitation; Counseling
MeSH Terms: conditions — Coronary Artery Disease; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interactive Voice Response Group (Experimental)
  Interventions: Behavioral: Interactive Voice Response
- Usual Care Group (No Intervention)

INTERVENTIONS:
Behavioral: Interactive Voice Response — The IVR group will receive a telephone call from the IVR system three, 14, 30, 90, 120 and 150 days after hospital discharge.
  Arms: Interactive Voice Response Group

SUMMARY:
A randomized control trial is planned to evaluate an interactive voice response (IVR) mediated follow-up and triage system, against usual care, to help smokers hospitalized with Coronary Heart Disease (CHD) to quit smoking. The investigators hypothesize that compared to usual care, participants in the IVR group will; a) have a significantly higher 7-day point prevalence abstinence rate at 26 and 52 weeks after hospital discharge, b) will have a higher rate of continuous abstinence at 26 and 52 weeks after hospital discharge, c) will use a greater number of proven effective interventions over time, and d) will develop greater self-efficacy with respect to smoking cessation, over time.

DETAILED DESCRIPTION:
Quitting smoking appears to be the single most effective intervention or treatment to reduce mortality in patients with Coronary Heart Disease (CHD). However, despite interventions, almost two-thirds of smokers resumed smoking in the year after hospitalization for CHD related illnesses; one-third resumed smoking within one month. A critical challenge for institution-level programs is how to provide consistent patient follow-up and linkage to community-based smoking cessation resources. Interactive voice response (IVR) technology has the potential to improve follow-up with smokers after hospitalization and to enhance triage to clinical support for smoking cessation. IVR uses natural language to place automated out-going calls that can pose questions regarding smoking status and progress with smoking cessation, that is then dropped into a database. A counselor is then able to link with the database and obtain information about the patient's smoking cessation needs and provide support as appropriate. A randomized control trial (RCT) is planned to evaluate whether an IVR system for follow-up and triage helps smokers hospitalized for CHD, quit smoking over 26- and 52-week follow-up periods. Participants are randomized into either a Usual Care or IVR group. Both groups will receive in-patient counseling and offer of nicotine replacement therapy. The IVR group will additionally receive a telephone call from the IVR system three, 14, 30, 60, 90, 120, and 150 days after hospital discharge. Variables that will be assessed at 26 and 52 weeks include: smoking status, both 7-day point-prevalent and continuous abstinence, as well as self-efficacy for smoking cessation, use of effective cessation resources and patient satisfaction (at 26 weeks).

ELIGIBILITY:
Inclusion Criteria:

1. Patient is currently a smoker (greater than 5 cigarettes per day in the month preceding admission);
2. Patient is 18 years of age and older;
3. Patient is admitted to the in-patient cardiology service at the University of Ottawa Heart Institute (UOHI) for: a) Acute Coronary Syndrome (includes patients admitted for unstable angina or acute myocardial infarction), b) Elective Percutaneous Coronary Intervention (PCI), c) Coronary Artery Bypass Graft (CABG) or d) diagnostic catheterization procedures related to CHD;
4. Patient has received automatic referral for smoking cessation counseling;
5. Patient is willing to provide informed consent

Exclusion Criteria:

1. Patient is unable to read and understand English;
2. Patient lives more than 1.5 hours from UOHI;
3. Patient is returning to referring institution/hospital

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 442 (Actual)
Dates: Start 2006-07; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Biochemically confirmed 7-day point prevalent smoking abstinence | 52 weeks

SECONDARY OUTCOMES:
Use of smoking cessation resources | 26 & 52 weeks
Self-efficacy in regards to smoking cessation | 26 & 52 weeks
Patient Satisfaction of the IVR system | 26 weeks
Continuous Abstinence since hospitalization | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Reid, PhD., Study Chair — University of Ottawa Heart Institute, Minto Prevention and Rehabilitation Centre; Andrew Pipe, C.M, MD, Principal Investigator — University of Ottawa Heart Institute, Minto Prevention and Rehabilitation Centre; Bonnie Quinlan, BSCN, Principal Investigator — University of Ottawa Heart Institute, Prevention and Rehabilitation Centre; Heather Sherrard, BSCN, MHA, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Reid RD, Aitken DA, Mullen KA, McDonnell L, Armstrong A, LeBlanc AG, Slovinec-D'Angelo M, Pipe AL. Automated Telephone Follow-up for Smoking Cessation in Smokers With Coronary Heart Disease: A Randomized Controlled Trial. Nicotine Tob Res. 2019 Jul 17;21(8):1051-1057. doi: 10.1093/ntr/nty108. PMID 29800420